CLINICAL TRIAL: NCT00105521
Title: A Double-Blind, Placebo-Controlled, Multicenter, Multinational Phase III Study to Evaluate the Safety and Efficacy of Sarizotan in Patients With Parkinson's Disease Suffering From Treatment-Associated Dyskinesia
Brief Title: Sarizotan in Participants With Parkinson's Disease Suffering From Treatment Associated Dyskinesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR 62225-019
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease; Dyskinesia
Keywords: Parkinson's Disease; Dyskinesia; Dyskinesia associated with dopaminergic treatment
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — sarizotan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive placebo matched to sarizotan tablet orally twice daily up to Week 12.
  Interventions: Drug: Placebo
- Sarizotan 2 milligrams per day (mg/day) (Experimental): Participants will receive sarizotan 2 milligrams (mg) per day (given in 2 divided daily doses) up to Week 12.
  Interventions: Drug: Sarizotan
- Sarizotan 4 mg/day (Experimental): Participants will receive sarizotan 4 mg/day (given in 2 divided daily doses) up to Week 12.
  Interventions: Drug: Sarizotan
- Sarizotan 10 mg/day (Experimental): Participants will receive sarizotan 10 mg/day (given in 2 divided daily doses) up to Week 12.
  Interventions: Drug: Sarizotan

INTERVENTIONS:
Drug: Sarizotan — Sarizotan will be administered twice daily.
  Arms: Sarizotan 10 mg/day; Sarizotan 2 milligrams per day (mg/day); Sarizotan 4 mg/day
Drug: Placebo — Placebo matching to sarizotan will be administered twice daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test multiple doses of sarizotan to establish a dose with maximal safety and efficacy for treating treatment associated dyskinesia in Parkinson's disease participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant is an out-patient
* The participant presents with a diagnosis of idiopathic Parkinson's disease
* Prior therapy with all registered Parkinsonian medication is allowed

Exclusion Criteria:

* (For female participants) The participant is pregnant or lactating
* The participant is participating in another clinical study or has done so within the past 30 days
* The participant has received neurosurgical intervention related to Parkinson's disease
* The participant has relevant renal impairment
* The participant has relevant hepatic impairment
* The participant is suffering from any dementia or psychiatric illness
* The participant has a history of allergic asthma

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2004-09-30 (Actual); Primary Completion 2006-03-31 (Actual); Study Completion 2006-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (28):
- United States (28):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Fayetteville, Arkansas
  - Fountain Valley, California
  - Los Angeles, California
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Ocala, Florida
  - Port Charlotte, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Columbia, Maryland
  - Boston, Massachusetts
  - Golden Valley, Minnesota
  - Omaha, Nebraska
  - Albany, New York
  - New York, New York
  - Syracuse, New York
  - Toledo, Ohio
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Upland, Pennsylvania
  - Dallas, Texas
  - Charlottesville, Virginia

REFERENCES:
- [Background] Goetz CG, Damier P, Hicking C, Laska E, Muller T, Olanow CW, Rascol O, Russ H. Sarizotan as a treatment for dyskinesias in Parkinson's disease: a double-blind placebo-controlled trial. Mov Disord. 2007 Jan 15;22(2):179-86. doi: 10.1002/mds.21226. PMID 17094088
- [Background] Goetz CG, Laska E, Hicking C, Damier P, Muller T, Nutt J, Warren Olanow C, Rascol O, Russ H. Placebo influences on dyskinesia in Parkinson's disease. Mov Disord. 2008 Apr 15;23(5):700-7. doi: 10.1002/mds.21897. PMID 18175337

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to sarizotan tablet orally twice daily up to Week 12.
- Sarizotan 2 mg/Day: Participants received sarizotan 2 milligrams per day (mg/day) (given in 2 divided daily doses) up to Week 12.
- Sarizotan 4 mg/Day: Participants received sarizotan 4 mg/day (given in 2 divided daily doses) up to Week 12.
- Sarizotan 10 mg/Day: Participants received sarizotan 10 mg/day (given in 2 divided daily doses) up to Week 12.
Period: Overall Study
Arm/Group | Placebo | Sarizotan 2 mg/Day | Sarizotan 4 mg/Day | Sarizotan 10 mg/Day
Started | 98 | 101 | 97 | 102
Completed | 83 | 90 | 80 | 85
Not Completed | 15 | 11 | 17 | 17
Not completed — Other | 1 | 1 | 2 | 0
Not completed — Adverse Event | 10 | 4 | 10 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 4
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 3 | 5 | 4 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Sarizotan 2 mg/Day: Participants received sarizotan 2 mg/day (given in 2 divided daily doses) up to Week 12.
- Total: Total of all reporting groups
Arm/Group | Placebo | Sarizotan 2 mg/Day | Sarizotan 4 mg/Day | Sarizotan 10 mg/Day | Total
Number analyzed (Participants) | 98 | 101 | 97 | 102 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.3) | 63.4 (9.2) | 63.2 (9.7) | 62.9 (8.7) | 63.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 47 | 37 | 45 | 177
  Male | 50 | 54 | 60 | 57 | 221

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Diary-Based On-Time Without Dyskinesia at Week 12
Description: On-time without dyskinesia was defined as a period (in hours) when the participant had no symptoms of off-time and was not asleep; also, participant had no difficulty in performing voluntary movements (that is, without dyskinesia). Off-time was defined as a period (in hours) when participant experienced increased parkinsonian symptoms (e.g. immobility or inability to move with ease). On-time was recorded by participant in a participant diary.
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat (ITT) population included all randomized participants who received at least one treatment dose and who had at least one follow-up visit assessment for an efficacy target outcome.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Placebo | Sarizotan 2 mg/Day | Sarizotan 4 mg/Day | Sarizotan 10 mg/Day
Number analyzed (Participants) | 95 | 96 | 93 | 97
hours/day | 1.6 (3.3) | 1.9 (3.8) | 1.7 (3.0) | 1.8 (3.1)

2. Secondary Outcome: Change From Baseline in Modified Abnormal Involuntary Movement Scale (AIMS) Score at Week 12
Description: Modified AIMS was a 7-item investigator-assessed scale to assess severity of dyskinesia. Each item was rated on a 0 (none) to 4 (severe) scale. Modified AIMS score was sum of the all item scores and ranged from 0 to 28, where higher score indicated increased severity. Modified AIMS score in resting state as well as with activity is reported.
Time Frame: Baseline, Week 12
Population: Modified ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sarizotan 2 mg/Day | Sarizotan 4 mg/Day | Sarizotan 10 mg/Day
Number analyzed (Participants) | 95 | 96 | 93 | 97
units on a scale
  Change at Week 12: Modified AIMS at Rest | -2.7 (5.7) | -3.0 (5.3) | -2.7 (4.1) | -3.7 (5.5)
  Change at Week 12: Modified AIMS with Activity | -3.0 (5.9) | -3.3 (5.6) | -3.0 (4.8) | -3.6 (6.0)

3. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Items 32 and 33 Composite Score at Week 12
Description: The UPDRS was an investigator-assessed rating tool to follow the longitudinal course of Parkinson's disease. Items 32 and 33 assessed duration of dyskinesia and disability due to dyskinesia, respectively. Both items were rated on a 0 to 4-point scale, where higher scores indicated higher duration of dyskinesia and more disability due to dyskinesia, respectively. The Items 32 and 33 composite score was sum of the individual item scores and ranged from 0 to 8, where higher score indicated more complications due to dyskinesia.
Time Frame: Baseline, Week 12
Population: Modified ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sarizotan 2 mg/Day | Sarizotan 4 mg/Day | Sarizotan 10 mg/Day
Number analyzed (Participants) | 95 | 96 | 93 | 97
units on a scale | -1.0 (1.4) | -1.4 (1.6) | -1.1 (1.4) | -1.3 (1.3)

4. Secondary Outcome: Change From Baseline in UPDRS Part III Total Score at Week 12
Description: The UPDRS was an investigator-assessed rating tool to follow the longitudinal course of Parkinson's disease. UPDRS Part III total score was the sum of the 27 answers (rated on 0 to 4-point scale) related to motor examination, and ranged from 0-108. Higher scores indicated worse motor function. Change from baseline in UPDRS Part III total score, assessed during on-time (time when the participant has no parkinsonian symptoms) as well as off-time (time when the patient experiences increased parkinsonian symptoms), is reported.
Time Frame: Baseline, Week 12
Population: modified ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sarizotan 2 mg/Day | Sarizotan 4 mg/Day | Sarizotan 10 mg/Day
Number analyzed (Participants) | 95 | 96 | 93 | 97
units on a scale
  Change at Week 12: UPDRS Part III On-Time | 0.3 (6.8) | -0.1 (6.4) | -0.1 (6.8) | -0.8 (7.1)
  Change at Week 12: UPDRS Part III Off-Time | -3.0 (8.7) | -1.1 (8.7) | -0.0 (7.6) | -1.8 (9.0)

ADVERSE EVENTS:
Description: Among serious adverse events (SAEs), only data for total # affected by any SAE is available. Due diligence was done and all potential information sources have been exhausted; no further information could be retrieved. Hence, for SAEs the preferred term is reported as "Not Available" and System Organ Class as "General Disorders".
Arm/Group | Placebo | Sarizotan 2 mg/Day | Sarizotan 4 mg/Day | Sarizotan 10 mg/Day
Serious Adverse Events (participants affected / at risk) | 5/98 | 8/101 | 7/97 | 2/102
Other Adverse Events (participants affected / at risk) | 81/98 | 78/101 | 75/97 | 85/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=98) | Sarizotan 2 mg/Day (N=101) | Sarizotan 4 mg/Day (N=97) | Sarizotan 10 mg/Day (N=102)
(General disorders) | 5 | 8 | 7 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=98) | Sarizotan 2 mg/Day (N=101) | Sarizotan 4 mg/Day (N=97) | Sarizotan 10 mg/Day (N=102)
Parkinsonism aggravated (Nervous system disorders) | 27 | 23 | 35 | 32
Dyskinesia aggravated (Musculoskeletal and connective tissue disorders) | 7 | 11 | 7 | 10
Nausea (Gastrointestinal disorders) | 6 | 6 | 7 | 13
Falls (Injury, poisoning and procedural complications) | 4 | 11 | 3 | 2
Tremor aggravated (Musculoskeletal and connective tissue disorders) | 5 | 7 | 1 | 6
Somnolence (Nervous system disorders) | 3 | 5 | 3 | 6
Fatigue (General disorders) | 5 | 6 | 3 | 2
Headache (Nervous system disorders) | 2 | 5 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4 | 5
Blood creatine protein kinase increased (Investigations) | 5 | 1 | 4 | 3
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 5 | 0 | 2 | 3

LIMITATIONS AND CAVEATS:
For SAEs, due diligence was done and all potential information sources have been exhausted, no further information could be retrieved apart from what is currently reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No